CLINICAL TRIAL: NCT02771535
Title: Long-term Efficacy of Metacognitive Training for Depression (D-MCT): a 3-year Follow up
Brief Title: Long-term Efficacy of Metacognitive Training for Depression (D-MCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1027/106
Record Dates: First submitted 2016-04-05; First posted 2016-05-13 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-MCT Group (Experimental): Metacognitive Training for Depression (D-MCT), 8 sessions (60min); twice a week over a period of 4 weeks. Metacognitive Training for depression (D-MCT) is a low-threshold, easy to administer group intervention. It aims at the reduction of depressive symptoms by changing cognitive biases; not only biases targeted in cognitive behavioral therapy but also those identified by basic research.
  Interventions: Behavioral: D-MCT
- Health Training Group (Active Comparator): Health Training Group (Walking/ Psychoeducation on health); 8 sessions (60min), twice a week over a period of 4 weeks
  Interventions: Behavioral: Health Training

INTERVENTIONS:
Behavioral: D-MCT — Metacognitive Training for Depression (D-MCT), 8 sessions (60min); twice a week over a period of 4 weeks. Metacognitive Training for depression (D-MCT) is a low-threshold, easy to administer group intervention. It aims at the reduction of depressive symptoms by changing cognitive biases; not only biases targeted in cognitive behavioral therapy but also those identified by basic research.
  Other Names: Metacognitive Training for Depression
  Arms: D-MCT Group
Behavioral: Health Training — Health Training Group (Walking/ Psychoeducation on health); 8 sessions (60min), twice a week over a period of 4 weeks
  Arms: Health Training Group

SUMMARY:
Aim of the current study is to investigate the long-term efficacy of Metacognitive Training for Depression (D-MCT) and to explore whether previously observed effects at the 6-month follow-up of a randomized, controlled, assessor-blind, parallel group trial are maintained at the 3-year follow-up.

DETAILED DESCRIPTION:
Dissemination of treatment for depression is still unsatisfying: every second patient does not receive, refuses, or is waiting for treatment. Moreover, with a drop-out rate of almost 25% in routine clinical practice, and a 54% relapse rate for treatment responders within the two years after treatment termination, improving treatment is necessary. Metacognitive Training for depression (D-MCT), a low threshold, easy to administer group intervention was designed to fill this gap. It aims at the reduction of depressive symptoms by changing cognitive biases; not only biases targeted in cognitive behavioral therapy but also those identified by basic research. It was positively evaluated with regard to feasibility and acceptance in a non-randomized pilot study. Moreover, efficacy of D-MCT was suggested in a randomized controlled trail (RCT) in comparison to an active control intervention (Jelinek et al., in press). In this trial patients with depressive disorder were completing a psychosomatic outpatient treatment program and were randomly assigned to either D-MCT or general health training. Severity of depression and cognitive biases were assessed at baseline (t0), post treatment (t1) and 6 months (t2) later by raters blind to diagnostic status. Intention-to-treat analyses demonstrated that at the end of treatment, as well as 6 months later, improvement in depression was significantly greater in the D-MCT relative to the health training group at medium effect sizes. A significantly greater number of patients in the D-MCT group were in remission at 6-month follow-up. Moreover, the decrease in cognitive biases and increase in psychological well-being/quality of life was larger in the D-MCT than the health training group over time. Aim of the current study is to investigate the long-term efficacy of D-MCT. For this purpose, an additional 3 year follow-up assessment (t3) is conducted. The Hamilton Depression Rating Scale (HDRS, 17-item version) total score serves as the primary outcome. Self-assessed depression, dysfunctional beliefs, self-esteem, quality of life, and ability to work serve as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria for the current study are:

* informed consent
* intention-to-treat-sample of the study Evaluation of Metacognitive Training for Depression (D-MKT) in psychosomatic rehabilitation, DRKS-ID: DRKS00007907 (see Jelinek et al., in press, Psychotherapy and Psychosomatics)
* age between 18 and 65 years
* diagnosis of a single episode or recurrent major depressive disorder (MDD) or dysthymia (verified by the MINI).

The exclusion criteria were:

* lifetime psychotic symptoms (i.e., hallucinations, delusions, or mania), suicidality (Suicidal Behaviors Questionnaire-Revised ≥ 7), intellectual disability (estimated IQ < 70).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 3 years from baseline (t0) to 3-year follow up (t3)
  Primary outcome is change on the Hamilton Depression Rating Scale (HDRS, 17-item version) from baseline to follow-up (t0 - t3)

SECONDARY OUTCOMES:
Self-assessed depression | 3 years from baseline (t0) to 3-year follow up (t3)
  Change in self-assessed depression as measured by the Beck-Depression Inventory (BDI) from baseline to follow-up (t0 to t3)
Dysfunctional beliefs | 3 years from baseline (t0) to 3-year follow up (t3)
  Change in dysfunctional beliefs as measured by the Dysfunctional Attitude Scale (DAS) from baseline to follow-up (t0 to t3)
Dysfunctional metacognitive beliefs | 3 years from baseline (t0) to 3-year follow up (t3)
  Change in metacognitive beliefs as measured by the Metacognitions Questionnaire (MCQ-30) from baseline to follow-up (t0 to t3)
Quality of life | 3 years from baseline (t0) to 3-year follow up (t3)
  Change in quality of life as measured by the World Health Organization Quality of Life Assessment (WHOQOL-BREF) from baseline to follow-up (t0 to t3)
Work status | at 3-year follow-up (t3)
  Work status (full or part-time employment, unemployed, house wife/husband, student, on sick leave, retired) at T3 assessment
Self-esteem | 3 years from baseline (t0) to 3-year follow up (t3)
  Change in self-esteem as measured by the Rosenberg Self-Esteem Scale (RSE) from from baseline to follow-up (t0 to t3)
Remission rate | at 3-year follow up (t3)
  Remission rate at T3 as measured by the Hamilton Depression Rating Scale (HDRS score ≤ 8)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Jelinek, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moritz S, Veckenstedt R, Andreou C, Bohn F, Hottenrott B, Leighton L, Kother U, Woodward TS, Treszl A, Menon M, Schneider BC, Pfueller U, Roesch-Ely D. Sustained and "sleeper" effects of group metacognitive training for schizophrenia: a randomized clinical trial. JAMA Psychiatry. 2014 Oct;71(10):1103-11. doi: 10.1001/jamapsychiatry.2014.1038. PMID 25103718
- [Background] Jelinek L, Hauschildt M, Wittekind CE, Schneider BC, Kriston L, Moritz S. Efficacy of Metacognitive Training for Depression: A Randomized Controlled Trial. Psychother Psychosom. 2016;85(4):231-4. doi: 10.1159/000443699. Epub 2016 May 27. No abstract available. PMID 27230865
- [Background] Jelinek L, Otte C, Arlt S, Hauschildt M: Denkverzerrungen erkennen und korrigieren: Eine Machbarkeitsstudie zum Metakognitiven Training bei Depression (D-MKT). [Identifying and correcting cognitive biases: A pilot study on the Metacognitive Training for Depression (D-MCT)]. Zeitschrift Für Psychiatr Psychol Und Psychother 61:1-8, 2013.